CLINICAL TRIAL: NCT07032753
Title: Neuromusculoskeletal Interface for Bionic Arms: A Randomized Crossover Study
Brief Title: Neuromusculoskeletal Interface for Bionic Arms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Integrum (Industry); Northwestern Memorial Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Levi Hargrove, Scientific Chair, Center for Bionic Medicine, Shirley Ryan Abilitylab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00223908; 1UG3NS127063-01A1 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Amputation; Amputation, Traumatic; Amputation, Surgical; Upper Limb Amputation Above Elbow (Injury)
Keywords: eOPRA for transhumeral amputees
MeSH Terms: conditions — Amputation, Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Investigators propose two randomized cross-over prospective clinical trials, in which each participant serves as his/her own control. Eight individuals with unilateral transhumeral amputations will undergo OI and TMR surgeries (Aim 2). After surgical healing and reinnervation of target muscles, subjects will participate in two clinical trials.
  Aim 3, subjects randomly assigned to either OPRA (surface EMG) or e-OPRA (implanted EMG) without sensory feedback. After training, subjects perform a set of outcome measures, then take the device home for 3 months with OPRA system (no EMG). They then return to the lab, complete the same outcome measures, then switch to the other system and repeat this protocol.
  Aim 4 follows the same study design, except that subjects will be randomly allocated to e-OPRA with or without sensory feedback, based on somatosensory maps collected in Aim 3. Subjects will use the same device for each condition and use pattern recognition to control the device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- OPRA implant system (Active Comparator): OPRA implant with surface EMG and myoelectric prosthesis system.
  Interventions: Device: OPRA
- eOPRA implant system (Experimental): eOPRA system with implanted EMG control and myoelectric prosthesis system.
  Interventions: Device: eOPRA
- eOPRA system without sensory feedback (Active Comparator): eOPRA implant system without sensory feedback and myoelectric prosthesis system.
  Interventions: Device: eOPRA without sensory feedback
- eOPRA system with sensory feedback (Experimental): eOPRA implant system with sensory feedback and myoelectric prosthesis system.
  Interventions: Device: eOPRA with sensory feedback

INTERVENTIONS:
Device: eOPRA — Electronic Osseoanchored Prostheses for the Rehabilitation of Amputees (e-OPRA) implant system for transhumeral amputees.
  Other Names: OPRA
  Arms: eOPRA implant system
Device: OPRA — Osseoanchored Prostheses for the Rehabilitation of Amputees (e-OPRA) implant system in individuals with transhumeral amputations
  Arms: OPRA implant system
Device: eOPRA with sensory feedback — Electronic Osseoanchored Prostheses for the Rehabilitation of Amputees (e-OPRA) implant system in individuals with transhumeral amputations with sensory feedback.
  Arms: eOPRA system with sensory feedback
Device: eOPRA without sensory feedback — Osseoanchored Prostheses for the Rehabilitation of Amputees (e-OPRA) implant system in individuals with transhumeral amputations without sensory feedback.
  Arms: eOPRA system without sensory feedback

SUMMARY:
The overall objective of this proposal is to perform a first-in-human home trial of the Electronic Osseoanchored Prostheses for the Rehabilitation of Amputees (e-OPRA) implant system in individuals with transhumeral amputations who have had Targeted Muscle Reinnervation (TMR) surgery and use a pattern recognition-controlled myoelectric prosthesis. The purpose of the study is to capture preliminary safety and effectiveness information on the e-OPRA device when used with the prosthetic systems. The investigators expect that the e-OPRA implant system will be safe and provide clinically and statistically significant improvements in control and comfort.

Specifically, the investigators hypothesize that the e-OPRA system will (1) allow for training of more functional prosthesis controllers, (2) provide more stable electromyographic (EMG) signals, reducing the need to recalibrate the prosthetic control system, and (3) be more comfortable, as it does not require a tethered arm-band to record surface EMG signals.

Phase 1: Perform TMR and e-OPRA surgeries in 8 persons with transhumeral amputations.

Phase 2: Perform a randomized cross-over study to compare the OPRA and e-OPRA system (without sensory feedback) in 8 transhumeral amputees who have received TMR.

Phase 3: Perform a randomized cross-over study to compare the e-OPRA system with and without sensory feedback in 8 transhumeral amputees who have received TMR.

DETAILED DESCRIPTION:
In the past decade, progress has been made in creating stronger, more capable prosthetic devices, with improved control. Similar improvements have been made in prosthesis suspension, which is a critically important factor in both comfort and function of a prosthetic device. While skin-fit suction sockets were considered the state of the art for many years, custom-rolled silicon and instrumented gel-liners are now becoming more common, as they provide improved comfort. However, these approaches still require use of an external socket worn on the residual limb.

The Osseoanchored Prostheses for the Rehabilitation of Amputees (OPRA) implant system (Integrum AB, Mölndal, Sweden) uses osseointegration (OI) (i.e., a metal implant is placed in the residual bone, which then grows into and integrates with the implant) to provide mechanical attachment of the prosthesis to the skeleton in the residual limb, thus eliminating the need for a socket.

However, obtaining electromyographic (EMG) control signals to enable myoelectric control of a prosthesis, whether it is attached through OI or a conventional socket, requires placement of surface electrodes over residual limb muscles, which has many practical limitations. Surface EMG signals are a complex blend of all local muscle activations and as such have low fidelity. It is difficult to isolate EMG signals from large surface muscles, and it is impossible to separate out signals from small or deep muscles. In addition, surface EMG signals are contaminated by several sources of noise, including ambient electromagnetic interference, motion artifact, and even electrocardiogram signals.

The limitations of surface electrodes may be overcome by surgically implanting the electrodes into the residual limb and placing them directly onto/into the tissue of the target muscle so that the EMG can be recorded directly at the source with improved signal to noise ratio and without disturbances from the external environment. Typically, such an approach would require skin-penetrating leads to convey the EMG signals from the implanted electrodes to the outside of the body to enable myoelectric prosthesis control, making it unsuitable as a permanent solution.

However, in the e-OPRA (electronic OPRA) device, the percutaneous interface of the OPRA Implant is utilized as a conduit for the wired communication between the inside and the outside of the body, eliminating the need for permanent skin penetrating leads and enabling a permanent solution for myoelectric prosthesis control using implanted electrodes. The e-OPRA system (which is not yet commercially available) developed by Integrum AB (Mölndal, Sweden), is built on decades of developing the OPRA system (which is commercially available).

In addition to electrodes placed on muscle tissue, the e-OPRA device also contains implanted electrodes which are placed directly around peripheral nerves, which may be used for neurostimulation to generate sensory feedback to the user. The e-OPRA device constitutes the only available technology that provides a bidirectional neuromusculoskeletal interface in whichimplanted electrodes both record EMG signals and provide peripheral nerve stimulation for sensory feedback.

Use of the e-OPRA device with the well-documented neuro-electronic capabilities of EMG control systems provides an alternative to traditional socket prostheses by establishing a load-bearing coupling between the patient's skeleton and prosthesis, including wired connection between muscles and nerves in the residual limb and the prosthesis.

The investigators first propose to secure an investigational device exemption (IDE) from the FDA to implant an e-OPRA system. After implantation of the device and targeted muscle reinnervation (TMR) surgery in eight subjects with transhumeral amputations, we propose two clinical trials to (i) compare comfort and function with implanted electrodes (e-OPRA) or surface electrodes (OPRA) and (ii) evaluate the effects of providing sensory feedback.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 70 years old
* Unilateral transhumeral level absence
* Candidate for a myoelectric prosthesis (can generate mV level electromyographic EMG signals as detected by surface electrodes).
* Candidate for TMR surgery as verified by surgical team
* Candidate for OPRA surgery as verified by surgical team
* English speaking

Exclusion Criteria:

* Significant new injury that would prevent use of a prosthesis: The ability to consistently wear a prosthesis and perform activities of daily living and specific performance tasks is necessary to evaluate the relative benefits of the interventions.
* Cognitive impairment sufficient to adversely affect understanding of, or compliance with, study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate usable, reliable data. The ability to obtain relevant user feedback through questionnaires and informal discussion adds significant value to this study. These cognitive impairments would be confirmed with the Mini-Mental State exam.
* Proximal nerve injury that would prevent TMR or sensory feedback
* Significant other comorbidity: Any other medical issues or injuries that would preclude completion of the study, use of the prostheses, or that would otherwise prevent acquisition of useable data by researchers. Examples include: injuries to the shoulder, cervical spine or sound side joint pain that would prohibit the participants from being able use a prosthesis. Medical conditions including unregulated high blood pressure or advanced heart disease that would exclude the participant as an appropriate surgical candidate.
* Individuals who smoke. This may interfere with the OPRA process from both bone healing and soft tissue standpoints.
* Individuals with active implants. This has been a restriction of prior FDA IDE to investigate e-OPRA.
* Pregnant women
* Non-English speaking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety related: Adverse Event reporting | Through study completion for each subject, on average 3 years.
  The number/percentage of subjects that successfully demonstrate the absence of any Serious Adverse Device Effects will be summarized along with a 95% confidence interval.
Effectiveness related: EMG Signal to Noise Ratio Testing | Month 11, Month 13, Month 16, Month 19, Month 22
  The investigators will quantify the signal-to-noise ratio (SNR) of EMG signals by comparing activity recorded during maximum voluntary contraction (MVC) to that recorded during rest. SNR will be calculated as the ratio of EMG signal power during contraction to the signal power during rest, using a standardized protocol consistent with our preliminary data. Each trial will consist of three repetitions of three-second MVCs, interleaved with three-second rest periods. From each repetition, the central 30% of both the contraction and rest epochs will be extracted to minimize edge effects and ensure steady-state measurement. These extracted segments will then be concatenated across repetitions to create two signal arrays: one representing active EMG and the other representing baseline noise. This metric will be used to evaluate the quality of EMG signal acquisition from both surface and implanted electrodes, and to ensure adequate fidelity for pattern recognition control.
Effectiveness related: Somatosensory Mapping | Month 11, Month 13, Month 16, Month 19, Month 22
  The projected field-the region on the phantom limb where an electrically evoked sensation is perceived-for each contact on the implanted spiral nerve cuff electrodes. This mapping will be performed at three stimulation levels: the detection threshold (the lowest amplitude at which a sensation is first perceived) and two suprathreshold amplitudes that fall within a safe, physiologically relevant, and comfortably perceptible range. These amplitudes will allow us to assess the size, intensity, and location of the perceived sensation change with increased stimulation. Projected fields will be recorded on a schematic of the hand and used to build a subject-specific somatotopic map. This map will inform which sensor signals (from the TASKA CX hand) are routed to which nerve cuff contacts during the sensory feedback phases of the study. Contact-response stability will be evaluated over time, as these experiments will be repeated each time outcomes are collected in the study.
Effectiveness related: EMG Signal to Noise Ratio Testing | Month 13, Month 16, Month19, Month 22
  The investigators will quantify the signal-to-noise ratio (SNR) of EMG signals by comparing activity recorded during maximum voluntary contraction (MVC) to that recorded during rest. SNR will be calculated as the ratio of EMG signal power during contraction to the signal power during rest, using a standardized protocol consistent with our preliminary data. Each trial will consist of three repetitions of three-second MVCs, interleaved with three-second rest periods. From each repetition, the central 30% of both the contraction and rest epochs will be extracted to minimize edge effects and ensure steady-state measurement. These extracted segments will then be concatenated across repetitions to create two signal arrays: one representing active EMG and the other representing baseline noise. This metric will be used to evaluate the quality of EMG signal acquisition from both surface and implanted electrodes, and to ensure adequate fidelity for pattern recognition control.
Effectiveness related: Somatosensory Mapping | Month 13, Month 16, Month19, Month 22
  The projected field-the region on the phantom limb where an electrically evoked sensation is perceived-for each contact on the implanted spiral nerve cuff electrodes. This mapping will be performed at three stimulation levels: the detection threshold (the lowest amplitude at which a sensation is first perceived) and two suprathreshold amplitudes that fall within a safe, physiologically relevant, and comfortably perceptible range. These amplitudes will allow us to assess the size, intensity, and location of the perceived sensation change with increased stimulation. Projected fields will be recorded on a schematic of the hand and used to build a subject-specific somatotopic map. This map will inform which sensor signals (from the TASKA CX hand) are routed to which nerve cuff contacts during the sensory feedback phases of the study. Contact-response stability will be evaluated over time, as these experiments will be repeated each time outcomes are collected in the study.

SECONDARY OUTCOMES:
Orthotics and Prosthetics User Survey-Upper Extremity Functional Status (OPUS-UEFS): | Month 11, Month 13, Month 16, Month 19, Month 22
  A 19-item, self-reported measure of an individual's ability to perform self-care and upper limb-based daily living tasks (e.g. button shirt, tie shoelaces) using a 5-point scale. Rasch analysis of the questionnaire ratings is used to calculate an overall measure of each subject's functional ability.
Jebsen Test of Hand Function | Month 11, Month 13, Month 16, Month 19, Month 22
  The Jebsen test includes seven subtests, including writing, turning over cards, picking up small objects, etc., in which the time taken to complete each subtask is recorded. The test has been validated for able-bodied subjects, but not for subjects with an amputation. The investigators have used this test previously for transhumeral and transradial amputees.
Clothespin Relocation Task | Month 11, Month 13, Month 16, Month 19, Month 22
  A test of prosthetic function that requires the user to move three clothespins from a vertical bar to a horizontal bar (thereby requiring use of the elbow, terminal device, and wrist rotator). This test has been in use by the Center for Bionic Medicine as a measure of prosthesis function for over a decade.
Modified Box and Block Test | Month 11, Month 13, Month 16, Month 19, Month 22
  This test involves counting the number of blocks a patient can move from one side of a box, over a barrier, to the other side of the box, usually in a 2-min test period. This test requires elbow and hand function.
Southhampton Hand Assessment Procedure (SHAP) | Month 11, Month 13, Month 16, Month 19, Month 22
  The SHAP is a clinically validated, objective (self-timed) test of unilateral hand function that can be used to evaluate functionality of passive, mechanical, or myoelectric hands without bias to type-and changes in control ability over time. Abstract objects (some light, some heavy) and activities of daily living that are classified into one (or more) of six hand grips are timed by the subject. Scores are compared to a normalized, able-bodied control score of 100 allowing assessment of functional control of the terminal device compared to an intact hand Although this test has not been validated in prosthesis users, it was recommended for use while undergoing validation for this population.
Assessment of Capacity for Myoelectric Control (ACMC) | Month 11, Month 13, Month 16, Month 19, Month 22
  The ACMC is an observational assessment tool that specifically measures the subject's ability to control a myoelectric hand and is the only validated test for subjects with an upper limb amputation. The ACMC uses a Rasch analysis of the subject's ability to control gripping, holding, releasing, and coordinating 30 items, and is scored on a four-point capability scale: 0, not capable; 1, sometimes capable; 2, capable on request; and 3, spontaneously capable. The prosthetic hand is used normally (i.e., in an active assist or passive support role). The test can detect small differences in ability to perform daily bimanual tasks and takes as little as 10-15 minutes to administer, although scoring takes significantly longer.
Patient-Specific Functional Scale (PSFS): | Month 11, Month 13, Month 16, Month 19, Month 22
  A questionnaire that asks patients to list up to five tasks they have difficulty with and rate the difficulty on an 11-point numerical scale. Difficulty ratings can be averaged for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Levi Hargrove, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan Abilitylab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided due to pending IDE.